CLINICAL TRIAL: NCT06051461
Title: Deciphering the Role of Dietary Fatty Acids on Extracellular Vesicles-mediated Intercellular Communication and Their Implication in Atherosclerosis and Metabolic Syndrome: a Multi-omics Approach to Precision Nutrition
Brief Title: Deciphering the Role of Dietary Fatty Acids on Extracellular Vesicles-mediated Intercellular Communication
Acronym: DIETEVOME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Spanish National Research Council (Other Government)
Responsible Party: Principal Investigator, Sergio Montserrat de la Paz, Professor, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: US
Record Dates: First submitted 2023-09-05; First posted 2023-09-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Metabolic Syndrome; Metabolic Disorder; Inflammation; Immune System and Related Disorders
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Metabolic Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolic Syndrome patients (Active Comparator)
  Interventions: Dietary Supplement: Oral lipid emulsions
- Healthy patients (Experimental)
  Interventions: Dietary Supplement: Oral lipid emulsions

INTERVENTIONS:
Dietary Supplement: Oral lipid emulsions — The oral lipid emulsions will contain water, sucrose, emulsifier, flavouring, and the corresponding fat (50 g/m2 of body surface area): milk cream (SFAs) or refined olive oil (MUFAs) with or without a dose of omega-3 PUFA, which will consist of 920 mg of EPA and 760 mg of DHA (ω3-LCPUFAs).

SUMMARY:
Dietary interventions have been consistently proposed as a part of a comprehensive strategy to lower the incidence and severity of atherosclerosis and coronary vascular disease. Excessive comsumption of fats enriched in saturated fatty acids (SFAs) is associated with an increased risk of atherosclerosis and other cardiovascular diseases (CVD). In contrasts, replacement of SFAs with monounsaturated fatty acids (MUFAs) and omega-3 long chain polyunsaturated fatty acids (ω3-LCPUFAs) has been reported to be inversely associated with risk of atherosclerosis. This is partly due to the ability of MUFAs (and ω3-LCPUFAs) to modulate lipoprotein composition, oxidation state, and consequently their functionality, among others. While most of the nutritional studies have focused on elucidating the mechanisms by which dietary fats affect lipoprotein particles, little or nothing is known about the regulatory effect of dietary fatty acids on extracellular vesicles (EVs). EVs are small phospholipid particles that convey molecular bioactive cargoes and play essential roles in intercellular communication and, hence, a multifaceted role in health and disease. For the first time, the purpose of this project is to establish whether the type of major fatty acids present on a diet (SFAs, MUFAs, or ω3-LCPUFAs) may alter the structure, cargo, and functionality of postprandial- and long-term-EVs. In the precision nutrition era, the investigators expect to offer a new insight on EVs and their relationship with dietary fatty acids through the following objectives: 1) To map changes in the lipidome, proteome, microtranscriptome, and functional properties of circulating EVs in healthy subjects and patients with metabolic syndrome (MetS) both at fasting and at postprandial state upon a challenge of a meal rich in SFAs, MUFAs, and ω3-LCPUFAs; 2) To analyse the contribution of postprandial triacylglyceride-rich lipoproteins (TRL) on EVs-mediated intercellular communication in a fatty acid-dependent manner; and 3) To determine the influence of diets rich in SFAs, MUFAs, and ω3-LCPUFAs on EVs in an animal model of atherosclerosis in the setting of MetS. Collectively, this project will provide fundamental insight into EV biology, and remarks the clinical and functional relevance and divergent consequences of dietary fatty acids in health and disease.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of metabolic syndrome

Exclusion Criteria:

* Allergy to dairy products
* Allergy to fish oil
* Vegetarian
* Tobacco smoker
* Current or recent (<4 wk) use of fish oil supplements or more than four times fish/week
* Received innoculations within 2 mo of starting the study or planned to during the study
* Donated or intended to donate blood from 2 mo before the study till 2 mo after the study
* Unstable body weight (no weight gain/loss >3 kg)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of cytokines in postprandial state | Up to 6 hours
  Pro-inflammatory and anti-inflammatory cytokines, including NFα, IL-1β, IL-6, IL-8, IL-10, ICAM-1, MCP-1, leptin, and adiponectin, in plasma will be measured using appropriate methods (EIA, ELISA, and/or Bioplex multiplex system) (mg/dl).
Evolution of inflammatory markers in postprandial state. [Time Frame: Up to 6 hours] | Up to 6 hours
  The acute phase protein (hsCRP), PAI-1, fibrinogen, transferrin, albumin, and myeloperoxidase (MPO) will be measured using appropriate methods (EIA, ELISA, and/or Bioplex multiplex system) (mg/dl).
Effect of EVs on gene expression in PBMCs | Up to 6 hours
  PBMCs will be isolated from the subjects' peripheral blood and treated with autologous circulating EVs for different times.
EV proteome | Up to 6 hours
  The quantification of exosome-derived proteins will be performed by nLC-MS/MS
EV lipidome | Up to 6 hours
  The analysis of intact lipids derived from exosomes will be performed by LC-MS
Ev microtranscriptome | Up to 6 hours
  Enriched RNA and miRNA derived from exosomes will be determined by Next Generation Sequencing (NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marquez-Paradas E, Gil-Sanchez G, Barrera-Chamorro L, Gonzalez-de la Rosa T, Miguel-Albarreal AD, Corell A, Montserrat-de la Paz S. Postprandial modulation of the surface profile and cellular origin of circulating extracellular vesicles by dietary fatty acid composition: A randomized crossover pilot study in young healthy adults. Clin Nutr. 2025 Dec 6;56:106539. doi: 10.1016/j.clnu.2025.11.023. Online ahead of print. PMID 41406627